CLINICAL TRIAL: NCT03153124
Title: Effects of Respiratory Muscle Training in Muscle Force, Functional Capacity and Quality of Life in Hemodialysis Patients
Brief Title: Respiratory Training in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, PHD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64024117.4.0000.5479
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Respiratory muscle strength; Renal insufficiency; Respiratory muscle training
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training (Experimental): - three months of intradialytic training of a physical therapy protocol with PowerBreath.
  Interventions: Other: Respiratory muscle training
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Respiratory muscle training — The intervention group will perform three months of intradialytic training of a physical therapy protocol with PowerBreath
  Arms: Respiratory muscle training

SUMMARY:
Patients with chronic kidney disease in hemodialysis have complex syndrome with diverse effects on cardiovascular, nervous, respiratory, musculoskeletal, immune and endocrine-metabolic systems. With regard to the musculoskeletal structure, there is progressive muscular loss with consequent increase in muscle weakness, limited resistance, exercise intolerance and fatigue, as well as functional and morphological abnormalities characteristic of uremic myopathy. Respiratory muscles are also affected as a result of uremic myopathy, with decreased strength and resistance. Objective: to analyze the impact of respiratory muscle training on muscle strength, functional capacity and quality of life of patients with chronic kidney disease on hemodialysis. Method: This is a prospective, randomized study involving 46 patients followed by the dialysis unit of a university hospital, over 18 years old, of both genders who underwent hemodialysis for more than six months and who signed the informed consent form. Patients will be allocated into two groups: respiratory muscle training with PowerBreath and control. All will be evaluated for demographic data, respiratory muscle strength, lung function, functional capacity and quality of life. The intervention group will perform three months of intradialytic training of a physical therapy protocol with PowerBreath. Both groups will be reevaluated after three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease undergoing hemodialysis for more than 6 months Both genders
* ged 18 years or older
* clinically stable
* who agreed to participate in the study by signing a free informed consent form

Exclusion Criteria:

* Patients with previous or current myoarticular or neurological disease;
* That require some urgent or elective surgical intervention during the protocol;
* Any cardiac decompensation such as arrhythmias, systolic blood pressure greater than 200mmHg or less than 60mmHg, diastolic blood pressure greater than 120mmHg or less than 40mmHg;
* Decompensated diabetes mellitus and acute systemic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Manovacuometry | Change from baseline in respiratory muscle force at 3 months
  RESPIRATORY MUSCLE FORCE
Spirometry | Change from baseline in Pulmonary Function at 3 months
  Pulmonary Function
Distance in six-minute walk test | change from baseline in distance at 3 months
  analysis of distance
Quality of life questionnaire | change from baseline in quality of life at 3 months
  Analysis of the quality of life
HRR1 | change from HR six minute walk test and seven minute
  heart rate recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Levey AS, Atkins R, Coresh J, Cohen EP, Collins AJ, Eckardt KU, Nahas ME, Jaber BL, Jadoul M, Levin A, Powe NR, Rossert J, Wheeler DC, Lameire N, Eknoyan G. Chronic kidney disease as a global public health problem: approaches and initiatives - a position statement from Kidney Disease Improving Global Outcomes. Kidney Int. 2007 Aug;72(3):247-59. doi: 10.1038/sj.ki.5002343. Epub 2007 Jun 13. PMID 17568785
- [Background] Kaltsatou A, Sakkas GK, Poulianiti KP, Koutedakis Y, Tepetes K, Christodoulidis G, Stefanidis I, Karatzaferi C. Uremic myopathy: is oxidative stress implicated in muscle dysfunction in uremia? Front Physiol. 2015 Mar 30;6:102. doi: 10.3389/fphys.2015.00102. eCollection 2015. PMID 25870564